CLINICAL TRIAL: NCT05957341
Title: Personalized Brain Functional Sectors(pBFS) Guided 20min Inter-session Interval rTMS Treatment for Major Depressive Disorder： a Randomized， Double-Blind， Sham-controlled Trial
Brief Title: pBFS Guided 20min Inter-session Interval rTMS Treatment for MDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPLMDDinterP
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Moderate Depression; Major Depressive Disorder; Severe Depression
Keywords: transcranial magnetic stimulation, rTMS; Major Depression, Moderate Depression, MDD; personalized neuromodulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active rTMS: 20min inter-session interval (Experimental): Three sessions of active rTMS would be delivered, with 1800 pulse/session and 20 min inter-session intervals.
  Interventions: Device: active rTMS: 20min inter-session interval
- active rTMS: 50min inter-session interval (Active Comparator): Three sessions of active rTMS would be delivered, with 1800 pulse/session and 50 min inter-session intervals.
  Interventions: Device: active rTMS: 50min inter-session interval
- sham rTMS: 20min inter-session interval (Sham Comparator): Three sessions of sham rTMS would be delivered, with 1800 pulse/session and 20 min inter-session intervals.
  Interventions: Device: sham rTMS: 20min inter-session interval
- sham rTMS: 50min inter-session interval (Sham Comparator): Three sessions of sham rTMS would be delivered, with 1800 pulse/session and 50 min inter-session intervals.
  Interventions: Device: sham rTMS: 50min inter-session interval

INTERVENTIONS:
Device: active rTMS: 20min inter-session interval — Participants will receive active TMS, with 3 sessions per day, 1800 pulses/session, and 20 min inter-session intervals, lasting for 21 days. Individualized targets will be generated using the pBFS method.
  Arms: active rTMS: 20min inter-session interval
Device: active rTMS: 50min inter-session interval — Participants will receive active TMS, with 3 sessions per day, 1800 pulses/session, and 50 min inter-session intervals, lasting for 21 days. Individualized targets will be generated using the pBFS method.
  Arms: active rTMS: 50min inter-session interval
Device: sham rTMS: 20min inter-session interval — The parameters in this group are the same as in the active rTMS: 20min inter-session interval group. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham rTMS: 20min inter-session interval
Device: sham rTMS: 50min inter-session interval — The parameters in this group are the same as in the active rTMS: 50min inter-session interval group. Stimulation was delivered by the same device as the active group fitted with a sham coil.
  Arms: sham rTMS: 50min inter-session interval

SUMMARY:
The investigators aim to explore the efficacy and safety of rTMS therapies with different intervals between sessions for treating patients with moderate to severe depression.

DETAILED DESCRIPTION:
FDA-approved intermittent theta burst stimulation (iTBS) for the treatment of depression disorder, reduces the duration of a single sequence treatment from 37 minutes to 3 minutes with traditional rTMS and gets the same antidepressant effect. Studies have shown that large doses and individualized target stimulation based on iTBS can improve the efficacy of rTMS and greatly save the time spent during patient treatment, but the effect of the interval between iTBS sessions on the efficacy is inconclusive. Previous studies on interval effect in rats based on iTBS have indirectly found that the waiting time between iTBS sessions of 50 to 90 minutes can maximize the cumulative effect of stimulation, so researchers mostly set the iTBS treatment interval to 50 minutes. However, most patients give up treatment because of the long wait time of 50 minutes, so it is urgent to explore the effect of short intervals of iTBS accepted easier by patients. In this study, we examined the intersession interval of 50 min vs. 20 min in the efficacy and safety of pBFS-guided TMS treatment in patients with moderate to severe depression.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 4:4:1:1 ratio to a 50-minute active rTMS group, a 20-minute active rTMS group, a 50-minute sham-control group, and a 20-minute sham-control group. And then all participants will undergo a 21-day rTMS treatment followed by two-week and four-week follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for the depression disorder without psychotic symptoms, and currently experiencing recurrence episodes.
* Hospitalized patients aged 18-65 years (inclusive), male or female.
* Total HAMD-17 score ≥20 before randomization.Total MADRS score ≥25 before randomization.
* Inadequate response to at least one antidepressant trial of adequate doses and duration.
* A stable antidepressant regimen for at least 4 weeks at a dose not lower than the prescribed range of drug use before randomization.
* Voluntarily participate in the trial and sign informed consent.

Exclusion Criteria:

* Meet diagnostic criteria for other mental disorders (such as schizophrenia, schizoaffective disorder, bipolar disorder, secondary depression, and so on);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, and light therapy within 3 months;
* Patients with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* Patients with serious heart, liver, kidney diseases, diabetes, and other serious physical diseases, causing symptoms and signs of brain abnormalities, or body failure;
* The female of childbearing potential plans to become pregnant during the trial, and the female who is pregnant or breastfeeding.
* Alcohol abuse or drugs abuse in the past 1 year;
* First-degree relatives have bipolar affective disorder. There is a significant risk of suicide (MADRS item 10 ≥ 5).
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Currently participating in clinical trials of other drugs or physical therapy (e.g. deep brain stimulation DBS, electroconvulsive therapy ECT, rTMS).
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
change in MADRS | Baseline and Day 21(immediate post-treatment)
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression

SECONDARY OUTCOMES:
change in MADRS | Baseline, Day 7, Day 14, Day 21, 2-week post-treatment, 4-week post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression
change in HAMD | Baseline, Day 7, Day 14, Day 21, 2-week post-treatment, 4-week post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The Ham-17 version consists of 17 items assessing mood, guilt, general somatic symptoms, work and activities, anxiety, and slowness of thought and speech. Each item is scored on a scale of 0 to 4, except for the somatic, sleep, and insight items which are scored 0 to 2. On the HAMD-17 there can be a total score of 52. Higher scores represent higher depression severity
change in QID_SR | Baseline, Day 7, Day 14, Day 21, 2-week post-treatment, 4-week post-treatment
  A provider-administered questionnaire was used to assess remission and recovery from depression. The 16-item QIDS_SR is a widely used self-report instrument covering depressive symptoms incorporating nine Diagnostic and Statistical Manual of Mental Disorder-IV (DSM-IV) diagnostic criteria for major depressive disorders. Each item is scored on a scale of 0 to 4. Higher scores represent higher depression severity.
change in HAMA | Baseline, Day 7, Day 14, Day 21, 2-week post-treatment, 4-week post-treatment
  The HAMA was one of the first rating scales developed to measure the severity of anxiety symptoms, and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory